CLINICAL TRIAL: NCT05516927
Title: The Sanderson Study: A Diagnostic Case-Control Study for the Development of Multiomics Blood Tests for Cancer Screening in a Real World Setting
Brief Title: The Sanderson Study: A Case Control Study for the Development of Multiomics Blood Tests for Cancer Screening
Status: Completed | Type: Observational
Sponsor: Freenome Holdings Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: The Sanderson Study/FRNM-006
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Newly-diagnosed Cancers; Non-cancer Controls
Keywords: Liquid Biopsy; Blood Test; Cancer Diagnostic; Genomics; Multiomics; Artificial Intelligence; Screening; Machine Learning; Freenome; Early Detection; Multicancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens will be de-identified and used to validate the performance characteristics of the Freenome test
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Cancer Group: * Collect Subject Data
  * Collect Blood Specimen
  Interventions: Diagnostic Test: Freenome Test
- Non-cancer Group: * Collect Subject Data
  * Collect Blood Specimen
  Interventions: Diagnostic Test: Freenome Test

INTERVENTIONS:
Diagnostic Test: Freenome Test — Participants who provide informed consent, meet the eligibility criteria and provide a blood sample for this study will be enrolled.

SUMMARY:
This protocol is a prospective, case-control multi-center diagnostic study to assess the sensitivity and specificity of blood-based screening tests for the early detection of multiple cancers.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥30 years within 30 days of enrollment
* Able and willing to provide blood samples per protocol
* Able to comprehend and willing to sign and date the informed consent and HIPAA
* Authorization documents
* Able and willing to allow existing health data to be utilized for study purposes

Key Exclusion Criteria:

* Any history of solid organ or bone marrow transplantation
* Any physical trauma or surgery requiring inpatient overnight hospitalization in the 30 days preceding enrollment
* Received a blood transfusion in the 30 days preceding enrollment
* A medical condition that, in the opinion of the Investigator, should preclude enrollment in the study
* Known to be pregnant
* Any therapy for cancer, including but not limited to surgery, chemotherapy, biologic therapy, immunotherapy, and/or radiation therapy in the 5 years preceding enrollment
* Participated or currently participating in a clinical research study in which an experimental medication has been administered during the 30 days preceding enrollment
* Participated or currently participating in another Freenome-sponsored clinical study
* For non-cancer groups: Any previous cancer diagnosis in the 5 years preceding enrollment; OR recurrence of the same primary cancer within any timeframe; OR concurrent diagnosis of multiple primary cancers within any timeframe
* For the cancer groups: Any previous cancer diagnosis in the 5 years preceding enrollment, apart from the current cancer diagnosis; OR recurrence of the same primary cancer within any timeframe; OR concurrent diagnosis of multiple primary cancers within any timeframe

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adults 30+ who have been newly diagnosed with cancer and treatment-naive
  * Adults 30+ without cancer
Sampling Method: Non-Probability Sample
Enrollment: 788 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Comparison of Blood Samples from Cancer Case and Non-cancer Control Participants | 12 months
  To compare blood samples from cancer case and non-cancer control subjects in order to develop and characterize blood-based multiomics tests in specific cancer types or in a combination of multiple cancers.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Crisp Regional Hospital, Cordele, Georgia
  - Silver Cross Hospital and Medical centers, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Margaret Mary, Batesville, Indiana
  - Henry Ford Health, Detroit, Michigan
  - Allina Health Cancer Institute, Minneapolis, Minnesota
  - Winona Health System, Winona, Minnesota
  - Carroll County Memorial Hospital, Carrollton, Missouri
  - Hannibal Regional Hospital, Hannibal, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Inspira Medical Center, Mullica Hill, New Jersey
  - St Joseph University, Paterson, New Jersey
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Bloomsburg Hospital, Bloomsburg, Pennsylvania
  - MUSC, Charleston, South Carolina
  - MacLeod Center for Cancer Treatment and Research, Florence, South Carolina
  - Elligo Health Research, Inc., Austin, Texas
  - INOVA, Fairfax, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No